CLINICAL TRIAL: NCT01787786
Title: Defining and Predicting the Ideal Infliximab Pharmacokinetic Profile Associated With Treatment Efficacy in Patients With Inflammatory Bowel Disease
Brief Title: Improving Treatment of Inflammatory Bowel Diseases Through Better Understanding Infliximab Drug and Antibody Levels
Acronym: OPTIMIZE
Status: Withdrawn | Type: Observational
Why Stopped: Unable to align the study questions with a complementary trial
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: RP1207
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Ulcerative Colitis; Optimal Use of infliximab
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Irritable Bowel Disease: Infliximab administered according to current FDA and EMS approved doses and intervals.

SUMMARY:
The purpose of this study is to develop a predictive model that will allow optimized dosing of infliximab for individual patients

DETAILED DESCRIPTION:
The use of pharmacokinetic analyses incorporating relevant determinants of the infliximab serum concentration can be used to develop a predictive model that will allow optimized dosing for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of CD or UC by usual criteria,
* moderate to severely active CD defined by a CDAI ≥ 220, with confirmed endoscopic activity (CDEIS ≥ 6) or moderate to severely active UC, defined by a Mayo Score ≥ 6, with a Mayo endoscopic subscore ≥ 2,
* a need for treatment with IFX for induction of remission as clinically indicated
* patients previously exposed to adalimumab and/or certolizumab who are naïve to infliximab will be allowed to participate.

Exclusion Criteria:

* perianal CD exclusively
* disease limited to the rectum in patients with UC (i.e., disease must extend ≥ 15 cm from the anal verge)
* patients with known antibodies to IFX (ADAs) at baseline
* a contraindication to infliximab therapy
* a contraindication to endoscopy
* an ostomy
* planned surgery
* evidence of severe or unstable hepatic, gastrointestinal, cardiovascular, respiratory, neurological, psychiatric, hematological or renal disease at the discretion of the investigator,
* Pregnancy or breastfeeding,
* treatment with any investigational drug in the past 30 days, or 5 half lives (whichever is longer).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with Crohn's Disease and 50 patients with Ulcerative Colitis from 10 centres (Canada, United States, Netherlands and Spain).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Analysis of Infliximab in patients with moderate to severely active ulcerative colitis and Crohn's Disease | 24 weeks
  The primary objective of this study is to define the PK profile of IFX in patients with CD and UC and to determine covariates influencing drug clearance.

SECONDARY OUTCOMES:
Quantification of relative strengths of individual determinants of infliximab pharmacokinetics | 24 weeks
  Assessment of potential interactions between these determinants.

OTHER OUTCOMES:
Identification of patients at baseline that would benefit from receiving higher does of infliximab due to accelerated drug clearance | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feagan, MD, Principal Investigator — Robarts Clinical Trials - Western University

REFERENCES:
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Reinisch W, Sandborn WJ, Rutgeerts P, Feagan BG, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Blank M, Lang Y, Johanns J, Colombel JF, Present D, Sands BE. Long-term infliximab maintenance therapy for ulcerative colitis: the ACT-1 and -2 extension studies. Inflamm Bowel Dis. 2012 Feb;18(2):201-11. doi: 10.1002/ibd.21697. Epub 2011 Apr 11. PMID 21484965
- [Background] Gisbert JP, Panes J. Loss of response and requirement of infliximab dose intensification in Crohn's disease: a review. Am J Gastroenterol. 2009 Mar;104(3):760-7. doi: 10.1038/ajg.2008.88. Epub 2009 Jan 27. PMID 19174781
- [Background] Maser EA, Villela R, Silverberg MS, Greenberg GR. Association of trough serum infliximab to clinical outcome after scheduled maintenance treatment for Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1248-54. doi: 10.1016/j.cgh.2006.06.025. Epub 2006 Aug 22. PMID 16931170